CLINICAL TRIAL: NCT02183285
Title: A 30 Day, Randomised, Double-blind, Double-dummy, Placebo-controlled, Multicentre Safety Trial to Evaluate the Tolerability Profile of Pharmaton PHL 00747 Soft Gelatine Capsules (Multivitamin, Multimineral + Omega-3 Fatty Acids) 1/Day p.o. and Pharmaton PHL 00747 Film-coated Tablets (Multivitamin, Multimineral Without Omega-3 Fatty Acids) 1/Day p.o. in Healthy, Young Female Subjects of Child-bearing Potential
Brief Title: Tolerability of Pharmaton PHL 00747 in Healthy, Young Female Subjects of Child-bearing Potential
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1209.1
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- PHL 00747 capsules (Experimental)
  Interventions: Dietary Supplement: Pharmaton PHL 00747 soft gelatine capsules; Dietary Supplement: Placebo film-coated tablets (fct)
- PHL 00747 tablets (Experimental)
  Interventions: Dietary Supplement: Pharmaton PHL 00747 film-coated tablets; Dietary Supplement: Placebo soft gelatine capsules
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo film-coated tablets (fct); Dietary Supplement: Placebo soft gelatine capsules

INTERVENTIONS:
Dietary Supplement: Pharmaton PHL 00747 soft gelatine capsules
  Arms: PHL 00747 capsules
Dietary Supplement: Pharmaton PHL 00747 film-coated tablets
  Arms: PHL 00747 tablets
Dietary Supplement: Placebo film-coated tablets (fct)
  Arms: PHL 00747 capsules; Placebo
Dietary Supplement: Placebo soft gelatine capsules
  Arms: PHL 00747 tablets; Placebo

SUMMARY:
To determine the tolerability and safety of Pharmaton PHL 00747 soft gelatine capsules and film-coated tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy female out-patients of child-bearing potential
* Ages ranging between 18 and 40 years
* Willing and able to give written informed consent in accordance to Good Clinical Practice (GCP) and local legislation prior to participation in the study

Exclusion Criteria:

* Contraindications to the use of any of the trial ingredients
* Known hypersensitivity to any of the ingredients
* Alcohol- or drug-addiction
* Currently participation in another trial, or has participated in a trial within the previous 30 days
* Known abnormal values of the laboratory tests (if detected after enrolment, subjects will continue the treatment provided there are no medical objections)
* Already taking other mult-vitamin products during the last 2 weeks

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2003-11; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Incidence of total drug-related adverse events assessed by the investigator | up to 30 days

SECONDARY OUTCOMES:
Incidence of all adverse events | up to 30 days
Changes from baseline in laboratory tests including Quick's test, activated partial thromboplastin time (aPTT) and cholesterol (total, HDL, LDL) | up to 44 days
Changes from baseline in vital signs (blood pressure and heart rate) | up to 30 days
Overall tolerability assessed by the subject and the investigator on a four-point rating scale | day 30
Overall acceptance of the medications (taste and after taste) by the subject on a four-point rating scale | day 30
Tolerability of the trial medications by the subject | up to 30 days